CLINICAL TRIAL: NCT06556173
Title: A Phase 2a, Single Site, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VTX3232 in Participants With Early-Stage Parkinson's Disease
Brief Title: Phase 2a Study of VTX3232 in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zomagen Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTX3232-203
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Parkinson Disease
Keywords: VTX3232; Idiopathic Parkinson's Disease; NLRP3 Inhibitor; Zomagen
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VTX3232 Dose A (Experimental)
  Interventions: Drug: VTX3232

INTERVENTIONS:
Drug: VTX3232 — Dose A

SUMMARY:
This is a study to understand if taking VTX3232 is safe in participants diagnosed with early stage idiopathic Parkinson's Disease (PD). Approximately 10 patients will take VTX3232 Dose A.

The study consists of a 30-day Screening Period (to see if a participant qualifies for the study), a 7-day Pre-Baseline Period, a 28-day Open Label Treatment period (a participant receives active Dose A), and a 14-day Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 40 years up to 80 years of age, inclusive, at the time of signing the informed consent, with BMI > 18.5 and < 32.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
* Diagnosis of idiopathic Parkinson's Disease between 0 and 60 months prior to screening.
* Score of 2 or less on Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV at screening.
* Have not received prior treatment with deep brain stimulation (DBS).
* If receiving treatment with symptomatic PD therapies, treatment must be stable. Note: The Medical Monitor should be contacted with any questions regarding concomitant therapies.
* A female participant is eligible if they are of nonchildbearing potential
* A male participant sexually active with a woman of child bearing potential is eligible if they agree to use contraception/barrier and refrain from donating sperm during the study and for at least 90 days after the last dose

Exclusion Criteria:

* Diagnosis of a Parkinsonian syndrome other than idiopathic Parkinson's Disease.
* A diagnosis of a significant central nervous system (CNS) disease other than Parkinson's disease; history of repeated head injury or traumatic brain injury; history of epilepsy or seizure disorder other than febrile seizures as a child.
* History of brain surgery.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) / Serious Adverse Event (SAE) Incidence Rate and Severity through study completion | Day 1 of treatment period through study completion, up to 6 weeks
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of VTX3232 in plasma and Cerebrospinal Fluid (CSF) at Day 28 | Day 1 of treatment period to Day 28 of treatment period
  Concentration of VTX3232 in plasma and CSF through 28 days of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Naik, PhD, Study Director — Zomagen Biosciences Ltd.
Locations (1):
- Local Site #840001, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided